CLINICAL TRIAL: NCT00616135
Title: A Clinical Evaluation Of Adipose Derived Regenerative Cells In The Treatment Of Patients With BrEast Deformities Post Segmental Breast ResecTion (Lumpectomy) With Or Without Radiation ThErapy. A Phase IV Post Market Study.
Brief Title: Study of Autologous Fat Enhanced w/ Regenerative Cells Transplanted to Reconstruct Breast Deformities After Lumpectomy
Acronym: RESTORE-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sean Gemmill, MS, RAC; Clinical Research Manager, Cytori Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESTORE-2
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Breast Neoplasms; Carcinoma, Ductal, Breast; Mammaplasty; Mastectomy, Segmental, Lumpectomy, Breast Reconstruction,
Keywords: Breast; Stem Cell; Adipose Derived Stem Cells; Adipose Derived Regenerative Cells; ADRC; Reconstructive Breast Surgery; Breast Reconstruction; Cancer; Carcinoma; Autologous fat transplantation; Autologous fat; Cosmetic breast deformities; Functional breast deformity; Lumpectomy; Segmental mastectomy; Quadrantectomy; breast conservation therapy
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ADRC-Enhanced Autologous Fat Transplant — Autologous fat harvested from the patient is enhanced with ADRCs derived from a portion of the harvested fat and transplanted into the breast(s) that have a volume deficit post lumpectomy. This is a single arm study with no control. All patients receive cell therapy.

SUMMARY:
A post-marketing study evaluating the transplantation of autologous fat augmented with Adipose Derived Regenerative Cells (ADRCs), in patients with functional and cosmetic breast deformities post segmental mastectomy or quadrantectomy (lumpectomy).

ELIGIBILITY:
Inclusion Criteria:

* Females with a history of T2N0M0 breast carcinoma (tumor ≤3 cm in largest dimension)
* Surgical or endoscopic segmental mastectomy or quadrantectomy (lumpectomy)
* Clean surgical margins
* No prosthesis in breast(s) to undergo treatment
* Ability to undergo lipoaspiration
* Last treatment for breast cancer ≥ 12 months prior to enrollment with absence of recurrence (patients on anti-estrogen adjuvant therapy are NOT excluded)
* No evidence of recurrence of cancer based on mammogram or breast exam prior to enrollment
* Objective signs of mild breast damage post Breast Conservation Therapy
* Type I Cosmetic Sequelae Classification
* A minimum of 1 cm of soft tissue (e.g. breast or fat) is available between the skin and chest wall at the recipient site
* A minimum of two-thirds of the breast is remaining post Breast Conservation Therapy
* No continuous adhesion of skin to bone >3 cm in diameter
* The volume and shape of the defect(s) must be conducive to correction during a single treatment session (maximum defect volume ≤150 mL in breast(s) to undergo treatment)

Exclusion Criteria:

* History of autoimmune disorder (e.g., Systemic Lupus Erythematosus [SLE])
* History of connective, metabolic or atrophic skin disease
* History of keloid scarring
* Chronic use (>7 consecutive days) of anticoagulants (such as aspirin) or NSAIDs within 15 days prior to enrollment
* Life expectancy ≤ 2 years
* Recurrence or active malignancy requiring radiation or surgical treatment ≤12 months prior to enrollment
* Presence of any other known malignancy
* Body Mass Index (BMI) >30
* Plan to undergo weight reduction surgery or foresee any significant weight changes during the study (defined as changes in BMI >5 compared to baseline
* Presence of contraindications to MRI

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Patient and physician satisfaction with functional and cosmetic results. Improvement in overall breast deformity measured at 12 months compared to baseline. | 12 months

SECONDARY OUTCOMES:
Change in breast volume and shape at 6 and 12 Months compared to baseline. Improvement in skin pigmentation abnormalities at 6 and 12 months compared to Baseline. Improvement in overall breast deformity at 6 Months compared to Baseline. | 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- Jules Bordet Institute of Cancer, Brussels, Belgium
- Università degli Studi di Firenze, Florence, Italy
- Spain (2):
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Instituto Valenciano Oncologia, Valencia
- Glasgow Royal Infirmary, Glasgow, Scotland, United Kingdom